CLINICAL TRIAL: NCT00748267
Title: Use of Pre-Operative Hypnosis to Reduce Post-Operative Pain and Anesthesia Related Side-Effects
Brief Title: Hypnosis in Reducing Pain and Other Side Effects in Women Undergoing Surgery for Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Michael Lew, City of Hope Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 08029; P30CA033572 (NIH); CHNMC-08029; CDR0000612523 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2008-09-05; First posted 2008-09-08 (Estimated); Last update posted 2011-03-07 (Estimated); Status verified 2011-03

CONDITIONS: Anxiety Disorder; Breast Cancer; Nausea and Vomiting; Pain
Keywords: anxiety disorder; pain; nausea and vomiting; breast cancer
MeSH Terms: conditions — Anxiety Disorders; Breast Neoplasms; Nausea; Vomiting; Pain | interventions — Hypnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: questionnaire administration
Procedure: hypnotherapy
Procedure: therapeutic conventional surgery

SUMMARY:
RATIONALE: Hypnosis may be effective in reducing pain and other side effects in women undergoing surgery for breast cancer.

PURPOSE: This clinical trial is studying how well hypnosis works in reducing pain and other side effects in women undergoing surgery for breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To test the feasibility of hypnosis as a pre-operative intervention for the reduction of surgical- and anesthesia-related symptoms in women undergoing lumpectomy with sentinel node biopsy, mastectomy, or mastectomy with lymph node dissection for locally recurrent breast cancer.
* To identify the physical symptoms (i.e., pain, nausea, and vomiting) and psychological symptoms (i.e., anxiety and distress) of patients undergoing hypnosis.
* To determine the length of stay in the Post Anesthesia Care Unit of patients undergoing adjunct hypnosis.
* To describe patient satisfaction with the hypnosis experience.
* To determine the effect size and calculate the sample needed for a randomized clinical trial using the results of this study.

OUTLINE: Patients undergo a scripted hypnotic intervention over 15 minutes within 1 hour prior to their planned surgical procedure. Upon completion of the intervention, patients proceed to the Preoperative Holding Area of the Surgery and Post Anesthesia Care Unit where they receive the standard of care for lumpectomy with sentinel node biopsy, mastectomy, or mastectomy with lymph node dissection.

Patients undergo collection of demographic information (i.e., age; gender; ethnicity; marital/partnered status; spiritual practice; family members in the home; stress management history; experience with the continuum of imagery/hypnosis practices; perceptions of concentration abilities; and favorite aromas, colors, and scenes from nature) at the time of consent using the Demographic Survey Questionnaire. They also undergo assessment of physical and psychological symptoms (i.e., pain, nausea, vomiting, anxiety, and generalized distress) at baseline (immediately prior to hypnotic induction) and after the intervention (prior to discharge from the Post Anesthesia Care Unit).

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of breast cancer
* Scheduled for breast surgery (i.e., lumpectomy with sentinel node biopsy, mastectomy, or mastectomy with lymph node dissection) with Dr. Garbaroglio
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* Able to speak and read English
* Able to follow instruction
* No uncontrolled major comorbid mental conditions (i.e., thought disorders)
* No uncontrolled major physical conditions (i.e., untreated congestive heart failure)

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No concurrent reconstruction surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-08; Primary Completion 2010-02 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Pain as measured by the Condensed Memorial Symptom Assessment Scale (CMSAS)-Modified at baseline (pre-intervention) and prior to discharge from the Post Anesthesia Care Unit
Nausea as measured by the CMSAS-Modified at baseline and prior to discharge from the Post Anesthesia Care Unit
Vomiting as measured by the CMSAS-Modified at baseline and prior to discharge from the Post Anesthesia Care Unit
Generalized distress as measured by the CMSAS-Modified at baseline and prior to discharge from the Post Anesthesia Care Unit
Anxiety as measured by the CMSAS-Modified at baseline and prior to discharge from the Post Anesthesia Care Unit
Surgical and anesthesia time
Recovery time
Medications
Levels of consciousness
Standard clinical measures of levels of anesthesia
Significant surgical events
Patient satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lew, MD, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (1):
- City of Hope Comprehensive Cancer Center, Duarte, California, United States